CLINICAL TRIAL: NCT07224048
Title: Helicobacter Pylori Screening and Treatment in the At-risk South Florida Community-AIM 2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Phathom Pharmaceuticals (Unknown); NRG Oncology (Other)
Responsible Party: Principal Investigator, Shria Kumar, Assistant Professor of Clinical Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20211207-AIM 2
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: H. Pylori Infection; Gastric Cancer; Gastritis H Pylori
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- At-Home Retesting Strategy (Experimental): Participants who test positive for H. pylori (HP), will receive a kit that contains a PYtest® 14C-Urea Breath Test (TriMed). Participants will complete the retest at-home at least 6 weeks after treatment. Study team will contact the participant to inquire about retesting and the post treatment survey. The kit will include an envelope, materials for the test, and a return form. PYtest® is a quantitative and non-invasive method for the diagnosis of HP. The test is conducted with the swallowing of a urea capsule. If gastric urease from HP is present, the urea is split to form carbon dioxide and ammonia. Ten minutes after the capsule is ingested, a breath sample is collected in a balloon. The balloon is tied and mailed along with the return form to be analyzed by an outside laboratory. The study team will call the participant to provide results. Those who retest positive will be instructed to seek treatment from their primary care provider.
  Interventions: Drug: PYTEST® 14C-Urea Capsule Breath Test (at Home)
- Standard Care Retesting Strategy (Active Comparator): Participants who test positive for H. pylori (HP), will complete their retest in-person with the study team. Study team will contact the participant to inquire about scheduling the retest and the post treatment survey. Retest will be completed in Don Soffer or at one of study's community sites. PYtest® is a urea breath test and is a quantitative and non-invasive method for the diagnosis of HP. The test is conducted with the participant swallowing a urea capsule. If gastric urease from HP is present, the urea is split to form carbon dioxide and ammonia. Ten minutes after the capsule is ingested by the participant, a breath sample is collected in a balloon. This liquid is analyzed on site by the liquid scintillation counter, by the study team. Those who test positive will be instructed to seek treatment for H. pylori infection.
  Interventions: Drug: PYTEST® 14C-Urea Capsule Breath Test (Standard Retesting In-Person)

INTERVENTIONS:
Drug: PYTEST® 14C-Urea Capsule Breath Test (at Home) — FDA-approved radiolabeled urea capsule used in the PYtest® 14C-Urea Breath Test for non-invasive detection of Helicobacter pylori. Participants ingest the capsule as part of the at-home retesting protocol. If H. pylori is present, gastric urease hydrolyzes the urea, producing radiolabeled carbon dioxide detectable in the breath sample. The capsule is provided in a self-administered kit assembled by the study team and returned to a TriMed-associated lab for analysis.
  Arms: At-Home Retesting Strategy
Drug: PYTEST® 14C-Urea Capsule Breath Test (Standard Retesting In-Person) — FDA-approved radiolabeled urea capsule used in the PYtest® 14C-Urea Breath Test for non-invasive detection of Helicobacter pylori. In the standard retesting arm, participants ingest the capsule scheduled in-person. Ten minutes after ingestion, a breath sample is collected by clinical staff using a mylar balloon. The sample is sealed, labeled, and sent to a TriMed-associated laboratory for analysis using a liquid scintillation counter. The test detects the presence of H. pylori by measuring radiolabeled carbon dioxide produced by bacterial urease activity. Results are communicated to participants by the study team, and those who test positive are advised to seek treatment from their primary care provider.
  Arms: Standard Care Retesting Strategy

SUMMARY:
H. pylori is an infection of the stomach that can cause chronic gastritis, gastric cancer and peptic ulcer disease. The goal of this study is to screen people for this infection and offer treatment for those who test positive for the infection. By treating those who are positive for H. pylori, there is an opportunity to prevent gastritis, peptic ulcer disease, and even gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants in Aim 1 that received a positive result for H. Pylori (HP) testing
* Participants are advised to only begin re-testing procedures in Aim 2 if they have finished the medication regimen for HP treatment at least 6 weeks ago

Exclusion Criteria:

* Pregnant women, those who are breastfeeding, or those who are planning to become pregnant/breastfeed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-11-06 (Estimated); Study Completion 2027-11-06 (Estimated)

PRIMARY OUTCOMES:
Standard vs At-Home Retesting for eradication | 6 weeks after completion of treatment
  Percent of participants who complete at-home retesting, compared to the percent of participants who complete standard retesting, with successful eradication defined as obtaining a negative test result upon retesting.

CONTACTS AND LOCATIONS:
Overall Officials: Shria Kumar, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No